CLINICAL TRIAL: NCT05638100
Title: Efficacy and Safety of Different Doses of Rivaroxaban in Elderly Chinese Patients With Nonvalvular Atrial Fibrillation
Acronym: ESDDRECPNAF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-LCYJ-PY-32
Record Dates: First submitted 2022-11-06; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rivaroxaban-H: elderly patients (≥75-year-old) with NVAF administered Rivaroxaban(20mg/15mg)
- Rivaroxaban-M: elderly patients (≥75-year-old) with NVAF administered Rivaroxaban(10mg)
- Rivaroxaban-L: elderly patients (≥75-year-old) with NVAF administered Rivaroxaban(7.5mg)

SUMMARY:
From January 2023 to December 2025, 300 elderly patients with nonvalvular atrial fibrillation in Drum Tower Hospital Affiliated to Medical Scholl of Nanjing University will be enrolled to compare the efficacy and safety of rivaroxaban-H, rivaroxaban-M and rivaroxaban-L dose in elderly patients after 24-month follow-up.

DETAILED DESCRIPTION:
To explore the appropriate dose of rivaroxaban to prevent stroke in elderly Chinese patients with nonvalvular atrial fibrillation in order to improve the effectiveness and safety of anticoagulation therapy. From January 2023 to December 2025, 300 elderly patients with nonvalvular atrial fibrillation in Drum Tower Hospital Affiliated to Medical Scholl of Nanjing University will be enrolled to compare the efficacy and safety of rivaroxaban-H, rivaroxaban-M and rivaroxaban-L dose in elderly patients after 24-month follow-up. The efficacy indexes include stroke, non-CNS systemic embolism, fatal stroke, transient ischemic attack and myocardial infarction, and the safety indexes include major bleeding, non-major clinically relevant bleeding, minor bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Age≥75 years
* Chinese patient: male or female
* Patients had to be diagnosed as nonvalvular atrial fibrillation (NVAF)

Exclusion Criteria:

* Patients with anemia (hemoglobin<100g/L), known human immunodeficiency virus infection, female patients who were pregnant or lactating and patients for whom warfarin was contraindicated, were also excluded
* Patients with calculated creatine clearance vulue<30ml/min
* Patients expected to chronically use a non-steroidal anti-inflammatory agent (except for external preparations) and those treated with a strong cytochrome P4503A4 inhibitor (eg, ketoconazole, clarithromycin, or protease inhibitors) or a strong cytochrome P450 3A4 inducer (eg, rifampicin) during the trial

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Chinese patients aged ≥75 years with nonvalvular atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of stroke, non-CNS systemic embolism, fatal stroke, transient ischemic attack,myocardial infarction | January 2023-December 2025
  collect the information of patients enrolled in this study suffered from stroke, non-CNS systemic embolism, fatal stroke, transient ischemic attack, myocardial infarction
incidence of major bleeding, non-major clinically relevant bleeding, minor bleeding events | January 2023-December 2025
  collect information of patients enrolled in this study suffered from major bleeding, non-major clinically relevant bleeding, minor bleeding events